CLINICAL TRIAL: NCT05061420
Title: A Phase 2 Non-randomized, Open-label, Multi-cohort, Multi-center Study Assessing the Clinical Benefit of SAR444245 (THOR-707) Combined With Other Anticancer Therapies for the Treatment of Participants With Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: A Study of SAR444245 Combined With Other Anticancer Therapies for the Treatment of Participants With HNSCC (Master Protocol) (Pegathor Head and Neck 204)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on strategic sponsor decision not driven by any safety concerns.
Sponsor: Sanofi (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT16903; U1111-1251-5073 (Registry Identifier: ICTRP); KEYNOTE-B75 (Other: Merck Sharp & Dohme LLC.); 2021-002105-99 (EudraCT Number)
Record Dates: First submitted 2021-09-21; First posted 2021-09-29 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort A1 (sub study 01) treatment- naïve (Experimental): Participants with HNSCC, who were treatment-naïve for R/M disease and have a PD-L1 Combined Positive Score (CPS) ≥1, received pembrolizumab followed by SAR444245. Both drugs administered by intravenous (IV) infusion on Day 1 of each 21-day treatment cycle for up to 35 cycles.
  Interventions: Drug: Pembrolizumab; Drug: SAR444245 (Thor-707)
- Cohort B1: (sub study 04) PD1/PD-L1 and platinum-based treatments (Experimental): Participants with HNSCC who received treatment with a PD1/PD-L1-based regimen & platinum-based regimen and have failed no more than 2 regimens for R/M disease, received pembrolizumab followed by SAR444244. Both drugs administered IV infusion on Day 1 of each 21-day treatment cycle for up to 35 cycles
  Interventions: Drug: Pembrolizumab; Drug: SAR444245 (Thor-707)
- Cohort B2: (sub study 05) cetuximab- naïve (Experimental): Participants with R/M HNSCC, who were cetuximab-naïve, have received treatment with a platinum-based regimen, and have failed no more than 2 regimens for R/M disease, received treatment with cetuximab followed by SAR444245. Cetuximab IV was given on days 1, 8, and 15 of each 21 day. SAR444245 was administered by IV infusion on Day 1 of each 21-day treatment cycle. Dosing of both drugs continued until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: SAR444245 (Thor-707); Drug: Cetuximab

INTERVENTIONS:
Drug: Pembrolizumab — Pharmaceutical Form: Concentration for solution for infusion Route of Administration: Intravenous Infusion
  Other Names: KEYTRUDA®
  Arms: Cohort A1 (sub study 01) treatment- naïve; Cohort B1: (sub study 04) PD1/PD-L1 and platinum-based treatments
Drug: SAR444245 (Thor-707) — Pharmaceutical Form: Concentrate for solution for infusion Route of Administration: Intravenous Infusion
Drug: Cetuximab — Pharmaceutical Form: Solution for infusion Route of Administration: Intravenous Infusion
  Other Names: ERBITUX®
  Arms: Cohort B2: (sub study 05) cetuximab- naïve

SUMMARY:
The study was a phase 2 multi-cohort, non-randomized, open-label, multi-center study assessing the clinical benefit of SAR444245 combined with other anticancer therapies for the treatment of participants aged 18 years and older with HNSCC. This study was structured as a master protocol for the investigation of SAR444245 with other anticancer therapies.

Substudy 1-Cohort A1 aimed to establish proof-of-concept that SAR444245 combined with the anti-PD1 antibody pembrolizumab, will result in a significant increase in the observed number of objective responses in trial participants with HNSCC who were treatment-naïve for recurrent and/or metastatic (R/M) disease.

Substudy 4-Cohort B1 aimed to establish proof-of-concept that SAR444245 combined with the anti-PD1 antibody pembrolizumab, will result in a significant increase in the observed number of objective responses in trial participants with HNSCC who have received treatment with PD1/PD-L1 and platinum-based regimen.

Substudy 5-Cohort B2 aimed to establish proof-of-concept that SAR444245 combined with cetuximab will result in a significant increase in the observed number of objective responses in trial participants with HNSCC previously treated with platinum-based regimen & cetuximab-naive after failure of no more than 2 regimens for recurrent and/or metastatic (R/M) disease.

DETAILED DESCRIPTION:
The duration of the study for an individual participant started from the signature of the main informed consent and included:

* a screening period of up to 28 days
* a treatment period [max 35 cycles {cohort A1 and B1} = 735 days or until PD {cohort B2}]; max 35 cycles for SAR444245 and pembrolizumab]
* an end-of-treatment visit at least approximately 30 days following the last administration of study drug (or until the participant received another anticancer therapy, whichever was earlier)
* and a follow-up visits 3 months after treatment discontinuation and every 3 months thereafter following, until disease progression, or initiation of another antitumor treatment, or death, whichever was earlier

ELIGIBILITY:
Inclusion Criteria:

-Participants were ≥ 18 years of age inclusive, at the time of signing the informed consent

* Histologically or cytologically confirmed diagnosis of R/M HNSCC that was considered not amenable to further therapy with curative intent. The eligible primary tumor locations were oropharynx, oral cavity, hypopharynx, and larynx (nasopharynx is excluded).
* Measurable disease.
* Baseline biopsy was submitted for all cohort A1 Core Phase participants.
* Baseline biopsy was submitted for all cohort B1, B2 Expansion Phase participants.
* Known HPV p16 status for oropharyngeal cancer.
* Participant agreed to follow protocol-specified contraception guidelines.

Exclusion Criteria:

-Eastern Cooperative Oncology Group (ECOG) performance status of ≥2

* Had received prior IL2-based anticancer treatment. -For participants in Cohort A1: Prior treatment with an agent (approved or investigational) that blocks the PD-1/PD-L1 pathway (participants who joined a study with an anti-PD-1/PD-L1 in the experimental arm but have written confirmation they have not received anti-PD-1/PD-L1 are allowed).
* For participants in Cohort B2: Prior treatment with cetuximab (prior cetuximab allowed if used for the treatment of locally advanced disease, with no progressive disease for at least 4 months from completion of prior cetuximab therapy).
* For participants in Cohort B2: Electrolytes (magnesium, calcium, potassium) outside the normal ranges.
* Participants under anti-hypertensive treatment who cannot temporarily (for at least 36 hours) withhold antihypertensive medications prior to each IMP dosing.
* Participants with baseline SpO2 ≤92% (without oxygen therapy).
* Comorbidity requiring corticosteroid therapy (>10 mg prednisone/day or equivalent) within 2 weeks of IMP initiation. Inhaled or topical steroids are permitted, provided that they were not for treatment of an autoimmune disorder. Participants who require a brief course of steroids (eg, as prophylaxis for imaging studies due to hypersensitivity to contrast agents) were not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (27):
- United States (5):
  - City of Hope- Site Number : 8400007, Duarte, California
  - University of Colorado- Site Number : 8400004, Aurora, Colorado
  - University of Michigan- Site Number : 8400008, Ann Arbor, Michigan
  - Thomas Jefferson University Hospital Site Number : 8400003, Philadelphia, Pennsylvania
  - Seattle Cancer Care Alliance Site Number : 8400006, Seattle, Washington
- Investigational Site Number : 0320001, Buenos Aires, Argentina
- Investigational Site Number : 1240001, Montreal, Quebec, Canada
- Chile (4):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520002, Temuco
- France (5):
  - Investigational Site Number : 2500003, Bordeaux
  - Investigational Site Number : 2500008, Lyon
  - Investigational Site Number : 2500006, Paris
  - Investigational Site Number : 2500002, Strasbourg
  - Investigational Site Number : 2500001, Villejuif
- Investigational Site Number : 2760004, Berlin, Germany
- Investigational Site Number : 3800003, Brescia, Italy
- Netherlands (2):
  - Investigational Site Number : 5280002, Amsterdam
  - Investigational Site Number : 5280001, Nijmegen
- South Korea (2):
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (4):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240004, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240005, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240003, Madrid, Madrid, Comunidad de
- Investigational Site Number : 1580003, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217701&parentIdentifier=ACT16903&attachmentIdentifier=ddd9335a-c3e0-44fa-ade2-3328e8518d41&fileName=rdct-act16903-16-1-9-sap-PDFA.pdf&versionIdentifier=
- See also: ACT16903 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25204&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 27 centers (corresponds to number of site which screened at least one participant) in 12 countries. Out of 91 participants who were screened from 08 October 2021 to 21 October 2022, a total of 59 participants were enrolled in the study and were assigned to 1 of the 3 cohorts (Cohorts A1, B1 and B2) based on their disease type.
Pre-assignment Details: The study was terminated based on strategic sponsor decision not driven by any safety concerns. Cohort A2 was not initiated and no participants were enrolled. Note: Reason for not completed = Reason for permanent full intervention discontinuation.
Groups:
- CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy: Participants with head and neck squamous cell carcinoma (HNSCC) who were treatment-naïve for recurrent and/or metastatic (R/M) disease with programmed cell death-ligand 1 (PD-L1) combined positive score (CPS) >=1 were included in this cohort. Participants received pegenzileukin 24 microgram per kilogram (mcg/kg) along with pembrolizumab 200 milligram (mg) via intravenous (IV) infusion every 3 weeks (q3w) on Day 1 of each cycle (each cycle is 21 days) (as first line [1L] therapy), until disease progression (PD), unacceptable adverse event (AE), other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy: Participants with R/M HNSCC previously treated with programmed cell death protein (PD1)/PD-L1-based regimen and platinum-based regimen after failure of no more than 2 regimens for R/M disease were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as second or third line [2/3L] therapy), until PD, unacceptable AE, other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy: Participants with R/M HNSCC previously treated with platinum-based regimen and cetuximab-naïve after failure of no more than 2 regimens for R/M disease were included in this cohort. Participants received pegenzileukin 24 mcg/kg q3w on Day 1 of each cycle along with cetuximab as an initial loading dose of 400 mg/square meter (m^2) on Cycle 1 Day 1 followed by 250 mg/m^2 starting via IV infusion once weekly from Cycle 1 Day 8 (each cycle is 21 days) (as 2/3L therapy) until PD.
Period: Overall Study
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
Started | 20 | 20 | 19
Completed | 1 | 2 | 1
Not Completed | 19 | 18 | 18
Not completed — Adverse event: Not related to Coronavirus Disease 2019 (COVID-19) | 4 | 3 | 3
Not completed — Progressive disease | 11 | 15 | 14
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Not related to COVID-19 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The exposed population included all participants who had given their informed consent and received at least one dose of study treatment (pegenzileukin or other anticancer therapies).
Groups:
- CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy: Participants with HNSCC who were treatment-naïve for R/M disease with PD-L1 CPS >=1 were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 1L therapy), until PD, unacceptable AE, other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy: Participants with R/M HNSCC previously treated with PD1/PD-L1-based regimen and platinum-based regimen after failure of no more than 2 regimens for R/M disease were included in this cohort. Participants received pegenzileukin 24 mcg/kg along with pembrolizumab 200 mg via IV infusion q3w on Day 1 of each cycle (each cycle is 21 days) (as 2/3L therapy), until PD, unacceptable AE, other full permanent discontinuation criteria was met or completion of Cycle 35.
- Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy: Participants with R/M HNSCC previously treated with platinum-based regimen and cetuximab-naïve after failure of no more than 2 regimens for R/M disease were included in this cohort. Participants received pegenzileukin 24 mcg/kg q3w on Day 1 of each cycle along with cetuximab as an initial loading dose of 400 mg/m^2 on Cycle 1 Day 1 followed by 250 mg/m^2 starting via IV infusion once weekly from Cycle 1 Day 8 (each cycle is 21 days) (as 2/3L therapy) until PD.
- Total: Total of all reporting groups
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy | Total
Number analyzed (Participants) | 20 | 20 | 19 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.4) | 61.9 (8.8) | 58.8 (11.4) | 59.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 4 | 10
  Male | 18 | 16 | 15 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 1 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 10 | 12 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 9 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cohort A1: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 millimeter (mm) (<1 centimeter [cm]). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to approximately 21 months
Population: The efficacy population included all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy
Number analyzed (Participants) | 20
percentage of participants | 25.0 [10.4 to 45.6]

2. Primary Outcome: Cohort B1: Objective Response Rate
Description: ORR was defined as the percentage of participants who had a confirmed CR or PR as per RECIST v 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to approximately 21 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy
Number analyzed (Participants) | 20
percentage of participants | 0 [0.0 to 13.9]

3. Primary Outcome: Cohort B2: Objective Response Rate
Description: as for outcome 2
Time Frame: From first dose of study treatment administration (Day 1) up to approximately 21 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
Number analyzed (Participants) | 19
percentage of participants | 15.8 [4.4 to 35.9]

4. Secondary Outcome: All Cohorts: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any AE that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened (according to the Investigator's opinion) or became serious during the TE period.
Time Frame: From first dose of study treatment administration (Day 1) up to 30 days post last dose of study treatment administration, up to approximately 28 months (Cohort A1), 27 months (Cohort B1) and 26 months (Cohort B2)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
Number analyzed (Participants) | 20 | 20 | 19
Participants
  TEAEs | 20 | 20 | 19
  TESAEs | 11 | 11 | 8

5. Secondary Outcome: All Cohorts: Time to Response (TTR)
Description: TTR was defined as the time from the date of first study treatment administration to the first tumor assessment at which the overall response was recorded as PR or CR that was subsequently confirmed as per RECIST v 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 27 months (Cohort A1), 26 months (Cohort B1) and 25 months (Cohort B2)
Population: The efficacy population included all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment. Only participants with confirmed CR or PR were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
Number analyzed (Participants) | 5 | 0 | 3
months | 4.1 [2 to 7] |  | 2.1 [2 to 15]

6. Secondary Outcome: All Cohorts: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first tumor assessment at which the overall response was recorded as CR or PR that was subsequently confirmed to the date of first documentation of objective PD before the initiation of any post-treatment anti-cancer therapy or death due to any cause, whichever occurred first, as per RECIST v 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study), in addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm (0.5 cm).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
Number analyzed (Participants) | 5 | 0 | 3
months | 5.0 [3.9 to NA] — NA indicates that the upper limit of 90% confidence interval (CI) was not estimable due to insufficient number of participants with events. |  | 4.2 [4.2 to NA] — NA indicates that the upper limit of 90% CI was not estimable due to insufficient number of participants with events.

7. Secondary Outcome: All Cohorts: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with clinical benefit (confirmed CR or PR as best overall response [BOR], or SD lasting at least 6 months), as per RECIST v 1.1. CR was defined as the disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10mm (<1 cm). PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. BOR was defined as the best response recorded from the start of the study treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
Number analyzed (Participants) | 20 | 20 | 19
percentage of participants | 30.0 [14.0 to 50.8] | 0 [0.0 to 13.9] | 21.1 [7.5 to 41.9]

8. Secondary Outcome: All Cohorts: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of first study treatment to the date of the first documentation of objective PD or death due to any cause, whichever occurred first, as per RECIST v 1.1. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study), in addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm (0.5 cm).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
Number analyzed (Participants) | 20 | 20 | 19
months | 3.7 [2.0 to 6.9] | 1.9 [1.8 to 2.0] | 4.0 [2.0 to 6.0]

9. Secondary Outcome: Plasma Concentration of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of plasma concentration of pegenzileukin.
Time Frame: Cycle 1 Day 2 (each cycle is 21 days)
Population: The pharmacokinetic (PK) population included all participants from exposed population with at least one PK concentration available after the first dose of study treatment.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
Number analyzed (Participants) | 14 | 19 | 16
nanograms per milliliter | 173.0 (34.6) | 173.7 (55.5) | 188.8 (48.3)

10. Secondary Outcome: All Cohorts: Number of Participants With Anti-Drug Antibodies (ADAs) Against Pegenzileukin
Description: Blood samples were collected at specified timepoints to assess the presence of ADAs against pegenzileukin. Treatment-emergent ADA was defined as at least one treatment-induced or treatment-boosted ADA. Treatment-induced ADA was defined as ADA that developed during the TE period and without pre-existing ADA (including participants without pre-treatment samples). Treatment-boosted ADA was defined as pre-existing ADA that was boosted during the TE period to a significant higher titer than the baseline. Number of participants with treatment-emergent ADA are presented.
Time Frame: as for outcome 4
Population: The ADA population included all participants from exposed population with at least one ADA result (positive, negative or inconclusive) after the first dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
Number analyzed (Participants) | 20 | 20 | 18
Participants | 2 | 3 | 2

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from first dose of study treatment administration (Day 1) up to 30 days post last dose of study treatment administration, up to approximately 28 months (Cohort A1), 27 months (Cohort B1) and 26 months (Cohort B2). All-cause mortality (deaths) were collected from first dose of study treatment administration (Day 1) to the end of follow-up for death for each participant, up to approximately 30 months.
Description: Analysis was performed on the exposed population.
Arm/Group | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy
All-Cause Mortality (participants affected / at risk) | 8/20 | 13/20 | 10/19
Serious Adverse Events (participants affected / at risk) | 11/20 | 11/20 | 8/19
Other Adverse Events (participants affected / at risk) | 20/20 | 18/20 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy (N=20) | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy (N=20) | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy (N=19)
Abscess Neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atypical Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytokine Release Syndrome (Immune system disorders) | 3 (7) | 5 (11) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Cardiac Event (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardio-Respiratory Arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Capillary Leak Syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastrostomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Device Occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CohortA1:R/M HNSCC Treatment-naïve for R/M Disease:Pegenzileukin 24mcg/kg+Pembrolizumab as 1LTherapy (N=20) | Cohort B1: R/M HNSCC: Pegenzileukin 24 mcg/kg + Pembrolizumab as 2/3L Therapy (N=20) | Cohort B2: R/M HNSCC: Pegenzileukin 24 mcg/kg + Cetuximab as 2/3L Therapy (N=19)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 4 (7)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 2 (4) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (2) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Cytokine Release Syndrome (Immune system disorders) | 5 (9) | 0 (0) | 2 (3)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0)
Cell Death (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Brain Fog (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 4 (7)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (4)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 2 (2) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (8)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 4 (5) | 7 (10)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (26) | 3 (3) | 8 (19)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Oral Dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Salivary Hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 5 (9)
Tongue Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (18) | 3 (4) | 4 (12)
Cellulite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (12)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (3)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (3) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 5 (5)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (3)
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Discharge (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 2 (5) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Adverse Drug Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 6 (12) | 2 (3) | 2 (2)
Chills (General disorders) | 1 (14) | 5 (5) | 3 (3)
Fatigue (General disorders) | 5 (6) | 6 (10) | 6 (9)
Feeling Hot (General disorders) | 4 (5) | 1 (1) | 1 (1)
Hyperpyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza Like Illness (General disorders) | 1 (2) | 3 (4) | 2 (4)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (2)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (36) | 7 (12) | 4 (5)
Xerosis (General disorders) | 0 (0) | 0 (0) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 4 (4) | 2 (2) | 1 (4)
Aspartate Aminotransferase Increased (Investigations) | 3 (3) | 1 (1) | 1 (4)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Calcium Decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood Magnesium Decreased (Investigations) | 0 (0) | 0 (0) | 1 (4)
Blood Phosphorus Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 4 (5)
Weight Increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 5 (23)

LIMITATIONS AND CAVEATS:
The study was terminated based on strategic sponsor decision not driven by any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT05061420/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT05061420/SAP_001.pdf